CLINICAL TRIAL: NCT05184842
Title: Metabolically Optimized, Non-cytotoxic Low Dose Weekly Decitabine/Venetoclax in MDS and AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: The V Foundation for Cancer Research (Other); Icahn School of Medicine at Mount Sinai (Other); Servier (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13466
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — venetoclax; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Decitabine/Venetoclax (Single Arm) (Experimental): Administration: Decitabine is reconstituted with 5 ml sterile water to facilitate subcutaneous administration. Decitaboine is given by subcutaneous injection. Venetoclax is taken as a tablet prepared by patients pharmacy. Venetoclax is given at a dose of 400 mg po once per week concurrently with the Decitabine dose (+/- 1 day allowed ).
  Interventions: Drug: Venetoclax; Drug: Decitabine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax 400 mg po on days 1, 8, 15 and 22 of each cycle (28-day cycle)
Drug: Decitabine — Decitabine 0.2 mg/kg subcutaneous (SQ) on days 2, 9, 16, 23 (for aggressive disease will add decitabine on days 3, 10, 17, 24)

SUMMARY:
Myeloid malignancies which include AML (acute myeloid leukemia) and MDS (myelodysplatic syndrome) are cancers of the bone marrow which lead to bone marrow failure. The bone marrow is the place or factory in the body where components of blood such as red cells, platelets and white cells are made. In bone marrow failure, the ability of the bone marrow to make these cells is decreased. The decreased bone marrow function is the result from abnormalities that develop in the malignant cells which prevent the normal maturation process by which bone marrow cells develop into red blood cells, white blood cells and platelets. The malignant cells in the bone marrow are not good at maturing to make the components of the blood that you need, they occupy space in the bone marrow and prevent the function of remaining normal bone marrow cells.

DNA is a chemical substance within cells that stores information needed for cell growth and cell behavior. One approach to treating the malignant cells is to give chemotherapy which damages DNA within these cells and causes their death. Unfortunately, such therapy has side-effects, since even normal cells can be affected by the treatment.

Decitabine is FDA approved for treatment of MDS and AML. Venetoclax is approved for AML in combination with Azacitidine for patients with AML or are over age 75 or unfit for chemotherapy. In this study, Decitabine and venetoclax will be administered using a low dose weekly schedule in an attempt to improve efficacy by decreasing the side effects often seen when these drugs are given at standard dosing.

DETAILED DESCRIPTION:
The combination of Azacitidine and venetoclax (Aza/Ven) is FDA approved for patients AML > 75 and/or unfit for induction chemotherapy. However, majority of patients receiving standard dosing of Aza/Ven require dose interruptions, treatment delays and dose reductions. In addition, Aza/ven has limited activity in various subgroups of myeloid malignancies such as P53 mutant MDS/AML.

In the initial safety and tolerability phase of the study, 33 patients will be enrolled on this study, accounting for need for replacement subjects to evaluate endpoints. In the second expansion phase of the study up to 91 patients (including patients from the 1st stage), will be enrolled to obtain additional safety, tolerability and preliminary efficacy of the low dose regimen in selected subsets of patients with myeloid malignancies. As treatment with Hypomethylating agents (HMAs) requires extended drug exposure for efficacy, patients who do not complete 12 weeks of therapy for reasons other than disease progression or those who do not complete therapy due to toxicity or those who screen fail and do not start therapy, will be replaced. Any patient who starts therapy will be evaluable for safety. In the absence of overt disease progression or dose limiting toxicity, patients would be anticipated to remain on treatment for at least 12 weeks. After 12 weeks, patient may continue therapy if felt to be experiencing clinical benefit.

The severe cytopenias encountered with Aza/ven is particularly challenging for patients with poor hematopoietic bone marrow reserve such as MDS and myelofibrosis (MF). Also some elderly patients with comorbidities cannot tolerate the prolonged cytopenias caused by Aza/ven. This pilot clinical trial will evaluate the tolerability of a non-cytotoxic regimen for patients with myeloid malignancies who either cannot tolerate or are not known to benefit from standard Aza/Ven dosing.

This will be a single arm, open label pilot study of weekly dosing of subcutaneous decitabine and venetoclax. Patients will be treated for a minimum of 12 weeks in the absence of clear evidence of progressive disease. Patients who have any response will be permitted to continue treatment until relapse or progression of disease.

Decitabine is given at a dose of 0.1-0.2 mg/kg/day for 1-2 days per week. All patients will receive at least one dose Decitabine every week. If decided by treating physician that the patient needs a more rapid debulking of high disease burden, a second dose can be added. If Decitabine is given twice a week, should preferably be given on two consecutive days.

Venetoclax is dosed at 400 mg by mouth one day a week a day prior to the first decitabine dose. If patients are taking another CYP3A4 inhibitor dose adjustments should be made as recommended by pharmacist for a goal dose of venetoclax of 400 mg.

If patient receives two days of decitabine a week, they still only take venetoclax on the day prior to the first dose of decitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of myelodysplastic syndrome (MDS), acute myeloid leukemia (AML) or myelodysplastic/myeloproliferative neoplasms (MDS/MPN) with a histopathologic diagnosis confirmed by hematopathology review
* Indication for therapy with potential sensitivity to hypomethylating agents (HMA) therapy, defined as prior published evidence of response to HMA
* Patients must be 18 years of age or older
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 3
* Patients must have adequate end organ function defined as.

  * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) < 4× the upper limit of normal (ULN)
  * Bilirubin ≤ 2× the ULN (upper limit of normal). If elevated bilirubin is due to impaired conjugation (e.g., Gilbert's disease or concomitant medication) or disease related hemolysis, then direct bilirubin ≤ 1.5× the ULN
  * As decitabine and venetoclax have little renal metabolism, and have proven safety even in dialysis patients, renal function with a creatinine clearance ≥30 mL/min or on dialysis is allowed
* Subjects must have the ability to understand and the willingness to sign a written informed consent document and complete study related procedures.

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Core binding factor AML who are candidates for chemotherapy
* Prior Treatment with azacitidine, decitabine or venetoclax
* No other disease directed therapy, save for hydroxyurea, including experimental or investigational drug therapy for 14 days prior to study entry
* Currently pregnant or breast-feeding. Females of childbearing potential (FOCBP) must have negative serum pregnancy test within 72 hours from treatment start. (NOTE: FOCBP is any biologic female, regardless of sexual or gender orientation, having undergone tubal ligation, or remaining celibate by choice, who has not undergone a documented hysterectomy or bilateral oophorectomy or has had a menses any time in the preceding 12 months (therefore not naturally post-menopausal for > 12 months)
* Uncontrolled intercurrent illness that could limit life expectancy or ability to complete study correlates. This includes, but is not limited to:

  1. Ongoing or active infection. As patients with myeloid malignancies are prone to infections, if patients are actively being treated with appropriate antibiotics or antifungal therapy with clinical evidence of infection control, then they will be considered eligible for study.
  2. Uncontrolled concurrent malignancy
  3. Congestive heart failure of xNew York Heart Association (NYHA) class III/IV. Patients with compensated heart failure are permitted
  4. Unstable angina pectoris
  5. New or unstable cardiac arrhythmia. Stable or controlled arrhythmias are permitted
  6. Decompensated liver cirrhosis (Child-Pugh score ≥12 or a Model for Enst-Stage Liver Disease (MELD) score ≥21
  7. Psychiatric illness/social situations that would limit compliance with study requirements
  8. Any other prior or ongoing condition, in the opinion of the investigator, that could adversely affect the safety of the patient or impair the assessment of study results
* Women of Child-Bearing Potential (WOCBP) and males that are unwilling to agree to use dual contraceptive measures (i.e., hormonal or barrier method of birth control; abstinence, condom) prior to study entry and for the duration of study participation. Should a female subject become pregnant or suspect she is pregnant while participating in this study, she should inform the treating physician immediately
* Sexually active male who is unwilling to use a condom when engaging in any sexual contact with a female with child-bearing potential, beginning at the screening visit and continuing until 4 weeks after taking the last dose of Decitabine/venetoclax
* Patients with uncontrolled active HIV infection, as this will further increase the risk for opportunistic infections. However, patients with HIV with undetectable viral load by polymerase chain reaction (PCR), without opportunistic infection, and on a stable regimen of antiretroviral therapy would be eligible
* Known allergy or hypersensitivity to any component of decitabine or venetoclax formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2027-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Goldfinger, MD, Principal Investigator — Montefiore Medical Center
Locations (3):
- United States (3):
  - University of California Davis Health (UC Davis Health), Sacramento, California
  - Montefiore Medical Center, The Bronx, New York
  - White Plains Hospital, White Plains, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldfinger M, Mantzaris I, Shastri A, Saunthararajah Y, Gritsman K, Sica RA, Kornblum N, Shah N, Levitz D, Rockwell B, Shapiro LC, Gupta R, Pradhan K, Xue X, Munoz A, Dhawan A, Fehn K, Comas M, Verceles JA, Jonas BA, Kambhampati S, Shi Y, Braunschweig I, Cooper DL, Konopleva M, Feldman EJ, Verma A. A weekly low-dose regimen of decitabine and venetoclax is efficacious and less myelotoxic in a racially diverse cohort. Blood. 2024 Nov 28;144(22):2360-2363. doi: 10.1182/blood.2024025834. PMID 39316768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2022 and September 2023, 31 patients were enrolled. Nearly half of the patients were from diverse racial and ethnic backgrounds reflecting the demographics of an inner-city hospital in the Bronx, New York City.
Pre-assignment Details: 31 patients were consented/enrolled and comprised the Primary Outcome Measure analysis. Enrollment in progress at the time of this submission. The Primary Outcome Measure has been met and Results are being reported for the 31 participants who comprised the Primary Outcome Measure.
Groups:
- Decitabine/Venetoclax (Single Arm): Administration: Decitabine is reconstituted with 5 ml sterile water to facilitate subcutaneous administration. Decitabine is given by subcutaneous injection. Venetoclax is taken as a tablet prepared by patients pharmacy. Venetoclax is given at a dose of 400 mg po once per week concurrently with the Decitabine dose (+/- 1 day allowed ).
  Venetoclax: Venetoclax 400 mg po on days 1, 8, 15 and 28 of each cycle (28day cycle)
  Decitabine: Decitabine 0.2 mg/kg subcutaneous (SQ) on days 2, 9, 16, 23 (for aggressive disease will add decitabine on days 3, 10, 17, 24)
Period: Overall Study
Arm/Group | Decitabine/Venetoclax (Single Arm)
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analyses for initial group of 31 patients who comprised the Primary Outcome Measure.
Groups:
- Decitabine/Venetoclax (Single Arm): Administration: Decitabine is reconstituted with 5 ml sterile water to facilitate subcutaneous administration. Decitabine is given by subcutaneous injection. Venetoclax is taken as a tablet prepared by patients pharmacy. Venetoclax is given at a dose of 400 mg po once per week concurrently with the Decitabine dose (+/- 1 day allowed ).
  Venetoclax: Venetoclax 400 mg po on days 1, 8, 15 and 28 of each cycle (28day cycle)
  Decitabine: Decitabine 0.2 mg/kg SQ (subcutaneous) on days 2, 9, 16, 23 (for aggressive disease will add decitabine on days 3, 10, 17, 24)
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 73 [52 to 87]
Age, Continuous [Median (Full Range); unit: years] — Age, Continuous data is summarized for patients in the Acute Myeloid Leukemia (AML) cohort. Population: 21 of the 31 patients were part of the AML cohort.
  years
    number analyzed (Participants) | 21
    (all) | 75 [62 to 83]
Age, Continuous [Median (Full Range); unit: years] — Age, Continuous data is summarized for patients in the higher risk Myelodysplastic Syndrome (HR-MDS) cohort. Population: 6 of the 31 patients were part of the HR-MDS cohort.
  years
    number analyzed (Participants) | 6
    (all) | 61.5 [52 to 87]
Age, Continuous [Median (Full Range); unit: years] — Age, Continuous data is summarized for patients in the 'Other' cohort. Population: 4 of the 31 patients were part of the 'Other' (non AML or non HR-MDS) cohort.
  years
    number analyzed (Participants) | 4
    (all) | 67.5 [62 to 70]
Age, Customized [Count of Participants; unit: Participants] — The number/percentage of patients who are < 75 years old and ≥75 years old at baseline is summarized.
  Participants
    > 75 years old | 10
    < 75 years old | 21
Age, Customized [Count of Participants; unit: Participants] — Age, Customized data is summarized for patients in the AML cohort. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    > 75 years old: number analyzed (Participants) | 21
    > 75 years old | 9
    < 75 years old: number analyzed (Participants) | 21
    < 75 years old | 12
Age, Customized [Count of Participants; unit: Participants] — Age, Customized data is summarized for patients in the HR-MDS cohort. Population: 6 of the 31 patients were part of the HR-MDS cohort.
  Participants
    > 75 years old: number analyzed (Participants) | 6
    > 75 years old | 1
    < 75 years old: number analyzed (Participants) | 6
    < 75 years old | 5
Age, Customized [Count of Participants; unit: Participants] — Age, Customized data is summarized for patients in the 'Other' (non AML or non HR-MDS) cohort. Population: 4 of the 31 patients were part of the 'Other' cohort.
  Participants
    > 75 years old: number analyzed (Participants) | 4
    > 75 years old | 0
    < 75 years old: number analyzed (Participants) | 4
    < 75 years old | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Sex (Female, Male) summarized for initial group of 31 patients who comprised the Primary Outcome Measure.
  Participants
    Female | 17
    Male | 14
Sex: Female, Male [Count of Participants; unit: Participants] — Sex (Female, Male) is summarized for patients in the Acute Myeloid Leukemia (AML) cohort. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    number analyzed (Participants) | 21
    Female | 11
    Male | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Sex (Female, Male) is summarized for patients in the higher risk Myelodysplastic Syndrome (HR-MDS) cohort. Population: 6 patients were part of the higher risk Myelodysplastic Syndrome (HR-MDS) cohort.
  Participants
    number analyzed (Participants) | 6
    Female | 4
    Male | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Sex (Female, Male) is summarized for patients in the 'Other' cohort. This cohort was inclusive of patients with MDS/myeloproliferative neoplasm, chronic myelomonocytic leukemia, and myelofibrosis. Population: 4 patients were part of the 'Other' cohort. This cohort was inclusive of patients with MDS/myeloproliferative neoplasm, chronic myelomonocytic leukemia, and myelofibrosis.
  Participants
    number analyzed (Participants) | 4
    Female | 2
    Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Black | 6
  Hispanic | 7
  Asian | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity, Customized data is summarized for patients in the Acute Myeloid Leukemia (AML) cohort. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    White: number analyzed (Participants) | 21
    White | 12
    Black: number analyzed (Participants) | 21
    Black | 4
    Hispanic: number analyzed (Participants) | 21
    Hispanic | 4
    Asian: number analyzed (Participants) | 21
    Asian | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity, Customized data is summarized for patients in the higher risk Myeloid Dysplastic Syndrome (HR-MDS) cohort. Population: 6 of the 31 patients were part of the HR-MDS cohort.
  Participants
    White: number analyzed (Participants) | 6
    White | 4
    Black: number analyzed (Participants) | 6
    Black | 1
    Hispanic: number analyzed (Participants) | 6
    Hispanic | 1
    Asian: number analyzed (Participants) | 6
    Asian | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity, Customized data is summarized for patients in the 'Other' cohort. Population: 4 of the 31 patients were part of the 'Other' cohort.
  Participants
    White: number analyzed (Participants) | 4
    White | 0
    Black: number analyzed (Participants) | 4
    Black | 1
    Hispanic: number analyzed (Participants) | 4
    Hispanic | 2
    Asian: number analyzed (Participants) | 4
    Asian | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
Eastern Clinical Oncology Group (ECOG) Performance Status (PS) Scale [Count of Participants; unit: Participants] — The ECOG PS scale is a standardized measure which describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. ECOG PS grades range from 0-5; however, for this study only patients with an ECOG PS grade ≤ 3 are eligible. Brief ECOG PS grading is as follows: 0=fully active; 1=restricted in strenuous activity; 2=restricted in work activity but ambulatory and capable of self-care; 3=capable of limited self-care. Higher scores indicate increasing levels of disability. The number of patients with each grade is summarized.
  Participants
    ECOG PS = 0 | 13
    ECOG PS = 1 | 14
    ECOG PS = 2 | 4
    ECOG PS = 3 | 0
ECOG PS Scale - AML Cohort [Count of Participants; unit: Participants] — ECOG PS scale scores were summarized for the AML cohort. ECOG PS scores describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. Grades range from 0-5. For this study only patients with an ECOG PS grade ≤ 3 are eligible. Brief ECOG PS grading is as follows: 0=fully active; 1=restricted in strenuous activity; 2=restricted in work activity but ambulatory and capable of self-care; 3=capable of limited self-care. Higher scores indicate increasing levels of disability. The number of AML patients with each grade is summarized. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    ECOG PS = 0: number analyzed (Participants) | 21
    ECOG PS = 0 | 7
    ECOG PS = 1: number analyzed (Participants) | 21
    ECOG PS = 1 | 10
    ECOG PS = 2: number analyzed (Participants) | 21
    ECOG PS = 2 | 4
    ECOG PS = 3: number analyzed (Participants) | 21
    ECOG PS = 3 | 0
ECOG PS Scale - HR-MDS Cohort [Count of Participants; unit: Participants] — ECOG PS scale scores were summarized for the HR-MDS cohort. ECOG PS scores describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. Grades range from 0-5. For this study only patients with an ECOG PS grade ≤ 3 are eligible. Brief ECOG PS grading is as follows: 0=fully active; 1=restricted in strenuous activity; 2=restricted in work activity but ambulatory and capable of self-care; 3=capable of limited self-care. Higher scores indicate increased levels of disability. Number of HR-MDS patients with each grade is summarized. Population: 6 of the 31 patients were part of the HR-MDS cohort.
  Participants
    ECOG PS = 0: number analyzed (Participants) | 6
    ECOG PS = 0 | 4
    ECOG PS = 1: number analyzed (Participants) | 6
    ECOG PS = 1 | 2
    ECOG PS = 2: number analyzed (Participants) | 6
    ECOG PS = 2 | 0
    ECOG PS = 3: number analyzed (Participants) | 6
    ECOG PS = 3 | 0
ECOG PS Scale - Other Cohort [Count of Participants; unit: Participants] — ECOG PS scale scores were summarized for the 'Other' cohort. ECOG PS scores describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. Grades range from 0-5. For this study only patients with an ECOG PS grade ≤ 3 are eligible. Brief ECOG PS grading is as follows: 0=fully active; 1=restricted in strenuous activity; 2=restricted in work activity but ambulatory and capable of self-care; 3=capable of limited self-care. Higher scores indicate increasing levels of disability. The number of patients with each grade is summarized. Population: 4 of the 31 patients were part of the 'Other' cohort.
  Participants
    ECOG PS = 0: number analyzed (Participants) | 4
    ECOG PS = 0 | 2
    ECOG PS = 1: number analyzed (Participants) | 4
    ECOG PS = 1 | 2
    ECOG PS = 2: number analyzed (Participants) | 4
    ECOG PS = 2 | 0
    ECOG PS = 3: number analyzed (Participants) | 4
    ECOG PS = 3 | 0
Somatic mutations [Count of Participants; unit: Participants] — Somatic mutations common in MDS and AML blood cancers were confirmed prior to treatment. Responses to standard dosing of Hypomethylating agents (HMAs) (i.e., decitabine or azacytidine)/venetoclax have been most robust in AML with NPM1, IDH1, IDH2, or DNMT3A mutations; with limited activity in patients with P53, RAS and RUNX1 mutations. Patients with certain mutations may receive concomitant inhibitors during the study at the discretion of the PI, as outlined in the protocol. The number/percentage of patients with each mutation is categorized by type.
  Participants
    IDH1 or IDH2 | 6
    NPM1 | 1
    FLT3 ITD | 2
    N/KRAS | 4
    TP53 | 11
Somatic mutations - AML Cohort [Count of Participants; unit: Participants] — Somatic mutations specific to AML were confirmed prior to treatment. Responses to standard dosing of HMA (decitabine or azacytidine)/venetoclax have been most robust in AML with NPM1, IDH1, IDH2, or DNMT3A mutations; with limited activity in patients with P53, RAS and RUNX1 mutations. Patients with certain mutations may receive concomitant inhibitors during the study at the discretion of the PI, as outlined in the protocol. The number/percentage of AML patients with each mutation is categorized by type. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    IDH1 or IDH2: number analyzed (Participants) | 21
    IDH1 or IDH2 | 6
    NPM1: number analyzed (Participants) | 21
    NPM1 | 1
    FLT3 ITD: number analyzed (Participants) | 21
    FLT3 ITD | 2
    N/KRAS: number analyzed (Participants) | 21
    N/KRAS | 4
    TP53: number analyzed (Participants) | 21
    TP53 | 5
Somatic Mutations - HR-MDS Cohort [Count of Participants; unit: Participants] — Somatic mutations specific to HR-MDS were confirmed prior to treatment. Responses to standard dosing of HMA (decitabine or azacytidine)/venetoclax have been most robust in AML with NPM1, IDH1, IDH2, or DNMT3A mutations; with limited activity in patients with P53, RAS and RUNX1 mutations. Patients with certain mutations may receive concomitant inhibitors during the study at the discretion of the PI, as outlined in the protocol. The number/percentage of HR-MDS patients with each mutation is categorized by type. Population: 6 of the 31 patients were part of the HR-MDS cohort.
  Participants
    IDH1 or IDH2: number analyzed (Participants) | 6
    IDH1 or IDH2 | 0
    NPM1: number analyzed (Participants) | 6
    NPM1 | 0
    FLT3 ITD: number analyzed (Participants) | 6
    FLT3 ITD | 0
    N/KRAS: number analyzed (Participants) | 6
    N/KRAS | 0
    TP53: number analyzed (Participants) | 6
    TP53 | 6
Baseline Transfusion Dependence [Count of Participants; unit: Participants] — Patients with advanced myeloid malignancies often require frequent clinical visits and CBC evaluation for supportive transfusions. The number/percentage of patients requiring either packed red blood cell (RBC) and/or platelet transfusions to manage MDS/AML symptoms at the start of a study or treatment is summarized.
  Participants | 18
Baseline Transfusion Dependence - AML Cohort [Count of Participants; unit: Participants] — Patients with advanced myeloid malignancies often require frequent clinical visits and complete blood count (CBC) evaluation for supportive transfusions. The number/percentage of AML patients requiring either packed red blood cell (RBC) and/or platelet transfusions to manage their symptoms at the start of a study or treatment is summarized. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    number analyzed (Participants) | 21
    (all) | 11
Baseline Transfusion Dependence - HR-MDS Cohort [Count of Participants; unit: Participants] — Patients with advanced myeloid malignancies often require frequent clinical visits and CBC evaluation for supportive transfusions. The number/percentage of HR-MDS patients requiring either packed red blood cell (RBC) and/or platelet transfusions to manage their symptoms at the start of a study or treatment is summarized. Population: 6 of the 31 patients were part of the HR-MDS cohort.
  Participants
    number analyzed (Participants) | 6
    (all) | 5
Baseline Transfusion Dependence - Other Cohort [Count of Participants; unit: Participants] — Patients with advanced myeloid malignancies often require frequent clinical visits and CBC evaluation for supportive transfusions. The number/percentage of patients in the 'Other' cohort requiring either packed red blood cell (RBC) and/or platelet transfusions to manage their symptoms at the start of a study or treatment is summarized. Population: 4 of the 31 patients were part of the 'Other' cohort.
  Participants
    number analyzed (Participants) | 4
    (all) | 2
Acute Myeloid Leukemia (AML) Type [Count of Participants; unit: Participants] — AML patients enrolled into the study were categorized as being of either de novo origin, or of Secondary or therapy-related AML (t-AML) origin. de novo AML arises spontaneously, while secondary AML develops from prior a hematologic disorder and t-AML develops as a complication of prior cytotoxic therapy. The number/percentage of patients within each category/type is summarized with Secondary and t-AML being grouped as a single category. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    de novo: number analyzed (Participants) | 21
    de novo | 15
    Secondary (or t-AML): number analyzed (Participants) | 21
    Secondary (or t-AML) | 6
Bone Marrow Blast Count [Count of Participants; unit: Participants] — In Myelodysplastic Syndromes (MDS), bone marrow blast counts are a key factor in diagnosis and risk stratification. The number/percentage of patients with bone marrow myeloblast counts < 30% and ≥30% was characterized prior to treatment to differentiate between high blast and low blast patients. A bone marrow myeloblast count in excess of 30% is a strong indicator of acute myeloid leukemia (AML) while patients with lower blast count AML (<30%) are able to access MDS therapy. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    <30%: number analyzed (Participants) | 21
    <30% | 13
    ≥30%: number analyzed (Participants) | 21
    ≥30% | 8
European Leukemia Net (ELN) Risk Stratification Criteria [Count of Participants; unit: Participants] — ELN (2022) genetic risk stratification criteria were used to stratify AML patients into 3 risk strata based on genetic abnormalities prior to treatment. The 3 strata are Favorable Risk, Intermediate Risk, and Adverse Risk. The number/percentage of participants within each strata is summarized. Population: 21 of the 31 patients were part of the AML cohort.
  Participants
    Adverse Risk: number analyzed (Participants) | 21
    Adverse Risk | 14
    Intermediate Risk: number analyzed (Participants) | 21
    Intermediate Risk | 6
    Favorable Risk: number analyzed (Participants) | 21
    Favorable Risk | 1
Revised International Prognostic Scoring System (IPSS-R) Risk Category [Count of Participants; unit: Participants] — IPSS-R, a validated prognostic scheme, was used to classify patients with higher risk Myelodysplastic Syndrome (HR-MDS) into 1 of 5 risk categories based on how fast the disease is likely to progress, with risk categories corresponding to factors associated with increased mortality and an increased likelihood of the disease becoming AML. The categories of IPSS-R are determined based on a risk score: Very low-risk: ≤1.5; Low-risk: >1.5-3; Intermediate-risk: >3-4.5; High-risk: >4.5-6 and Very high-risk: >6. The number/percentage of HR-MDS patients within each category at baseline is summarized. Population: 6 of the 31 patients were part of the HR-MDS cohort.
  Participants
    Very low-risk: ≤1.5: number analyzed (Participants) | 6
    Very low-risk: ≤1.5 | 0
    Low-risk: 1.5 - 3: number analyzed (Participants) | 6
    Low-risk: 1.5 - 3 | 0
    Intermediate-risk: 3 - 4.5: number analyzed (Participants) | 6
    Intermediate-risk: 3 - 4.5 | 0
    High-risk: 4.5 - 6: number analyzed (Participants) | 6
    High-risk: 4.5 - 6 | 1
    Very high-risk: >6: number analyzed (Participants) | 6
    Very high-risk: >6 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Able to Continue on Treatment Without Dose Interruptions or Delays
Description: The percentage of participants who are able to continue on treatment without dose interruptions or delays was defined as not having to delay or interrupt treatment due to toxicity or intolerability for more than two weeks during the 12-week induction period.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 31
Participants
  Patients able to continue treatment during induction period without dose interruptions or delays | 28
  Patients who missed one or more doses during induction period | 3
  Patients requiring dose reduction(s) during induction period | 0

2. Secondary Outcome: Percentage of Participants With Complete Remission (CR) and Complete Remission With Incomplete Hematologic Recovery (CRi)
Description: Percentage of participants with CR + CRi will be calculated based on current International Working Group (IWG) criteria. CR is defined as absolute neutrophil count (ANC) > 1000/microliter (mcL), platelets > 100,000/mcL, red cell transfusion independence, and bone marrow with < 5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophils of ≤ 1000/mcL or platelets ≤ 100,000/mcL.
Time Frame: Up to 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Event-free Survival (EFS)
Description: EFS will be defined as the number of days from randomization to the date of progressive disease, relapse from CR or CRi, treatment failure or death from any cause.
Time Frame: Up to 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Complete Remission or Complete Remission With Partial Hematologic Recovery Rate (CR+CRh)
Description: A response of CRh is defined as Bone marrow with <5% blasts, peripheral blood neutrophil count >0.5*10^3/mcL and peripheral blood platelet count >0.5*10^5/mcL.
Time Frame: 3 months
Reporting Status: Not Posted

5. Secondary Outcome: Post Baseline Transfusion Independence Rate
Description: Transfusion Independence is defined as a period of 56 days with no transfusion between first dose of study drug and the last dose of study drug + 30 days. The rate of conversion for red blood cells (RBC) and platelets is defined as percentage of participants being post-baseline transfusion independent from baseline transfusion dependence.
Time Frame: Up to 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Hospitalization
Description: Rate of hospitalization will be defined as any hospitalization for complication related to myeloid malignancy or treatment. Initial admission for diagnosis or initiation of therapy will not be considered an event. For purposes of this study the rate of hospitalization will be defined as a percentage of participants who meet these criteria.
Time Frame: Up to 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Infection Rate Requiring Hospitalization
Description: Infection rate requiring hospitalization will be defined as being hospitalized due to a diagnosed infection or sepsis. For purposes of this study infection rate will be summarized as the percentage of patients who are diagnosed to have an infection or sepsis.
Time Frame: Up to 12 months
Reporting Status: Not Posted

8. Post Hoc Outcome: Overall Survival (OS) in AML Patients
Description: Median OS is reported in patients with AML at the time of censoring of data for the Primary Outcome analysis. For purposes of this study, OS refers to the duration of time from treatment initiation until a patient's death from any cause.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 21 patients who comprised the Primary Outcome analysis were part of the AML cohort.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Decitabine/Venetoclax (Single Arm): Administration: Decitabine is reconstituted with 5 ml sterile water to facilitate subcutaneous administration. Decitabine is given by subcutaneous injection. Venetoclax is taken as a tablet prepared by patients pharmacy. Venetoclax is given at a dose of 400 mg po once per week concurrently with the Decitabine dose (+/- 1 day allowed ).
  Venetoclax: Venetoclax 400 mg po on days 1, 8, 15 and 22 of each cycle (28-day cycle)
  Decitabine: Decitabine 0.2 mg/kg SQ (subcutaneous) on days 2, 9, 16, 23 (for aggressive disease will add decitabine on days 3, 10, 17, 24)
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 21
months | 16.1 [11.3 to NA] — An upper limit for the 95% Confidence Interval was unable to be reached for OS due to ongoing survival in some AML patients at the time of cutoff for data analysis (i.e., ~21 months).

9. Post Hoc Outcome: Overall Survival in HR-MDS Patients
Description: Median OS is reported in patients with HR-MDS at the time of censoring of data for the Primary Outcome analysis. For purposes of this study, OS refers to the duration of time from treatment initiation until a patient's death from any cause.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 6 patients who comprised the Primary Outcome analysis were part of the HR-MDS cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 6
months | 9.6 [8.5 to NA] — An upper limit for the 95% Confidence Interval was unable to be reached due for OS to ongoing survival in some HR-MDS patients at the time of cutoff for data analysis (i.e., ~21 months).

10. Post Hoc Outcome: Overall Response Rate (ORR) in Patients With AML by Intention-to-treat (ITT) Analysis
Description: ORR in patients with AML was determined by ITT analysis. ORR was defined by summarizing and calculating the number/percentage of patients with CR + CRi + Morphologic Leukemia-free State (MLFS), based on European LeukemiaNet (ELN) criteria. CR is defined as absolute neutrophil count (ANC) > 1000/microliter (mcL), platelets > 100,000/mcL, red cell transfusion independence, and bone marrow with < 5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophils of ≤ 1000/mcL or platelets ≤ 100,000/mcL. MLFS is defined as bone marrow blasts <5%; absence of blasts with Auer rods; and absence of extramedullary disease; no hematologic recovery required. Patients who have any response will be permitted to continue treatment until relapse or progression of disease. Results are summarized using basic descriptive statistics.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 21 patients who comprised the Primary Outcome analysis were part of the AML cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 21
Participants | 12

11. Post Hoc Outcome: Best Overall Response in Patients With AML Based on ITT Analysis
Description: Best Overall Response was determined in patients with AML who were analyzed by ITT analysis. The number/percentage of patients with Complete Remission (CR), Complete Remission with incomplete hematologic recovery (CRi), Morphologic Leukemia-free State (MLFS), and No Response is summarized based on ELN criteria summarized in corresponding Outcome Measures.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 21 patients who comprised the Primary Outcome analysis were part of the AML cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 21
Participants
  CR | 10
  CRi | 1
  MLFS | 1
  No Response | 9

12. Post Hoc Outcome: Overall Response Rate in Patients With AML by Intention-to-treat Per Protocol (ITT-PP) Analysis
Description: ORR in patients with AML was also determined by ITT-PP analysis. ORR was defined by summarizing and calculating the number/percentage of patients with CR + CRi + Morphologic Leukemia-free State (MLFS), based on European LeukemiaNet (ELN) criteria. CR is defined as absolute neutrophil count (ANC) > 1000/microliter (mcL), platelets > 100,000/mcL, red cell transfusion independence, and bone marrow with < 5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophils of ≤ 1000/mcL or platelets ≤ 100,000/mcL. MLFS is defined as bone marrow blasts <5%; absence of blasts with Auer rods; and absence of extramedullary disease; no hematologic recovery required. Patients who have any response will be permitted to continue treatment until relapse or progression of disease. Results are summarized using basic descriptive statistics.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 21 patients who comprised the Primary Outcome analysis were part of the AML cohort. Results for 2 of the 21 patients were not evaluable by ITT-PP analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 19
Participants | 12

13. Post Hoc Outcome: Best Overall Response in Patients With AML Based on ITT-PP Analysis
Description: Best Overall Response was also determined in patients with AML who were analyzed by ITT-PP analysis. The number/percentage of patients with Complete Remission (CR), Complete Remission with incomplete hematologic recovery (CRi), Morphologic Leukemia-free State (MLFS), and No Response is summarized based on ELN criteria summarized in corresponding Outcome Measures.
Time Frame: At the time of censoring of data, up to ~21 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 19
Participants
  CR | 10
  CRi | 1
  MLFS | 1
  No Response | 7

14. Post Hoc Outcome: Overall Response Rate in Patients With HR-MDS
Description: ORR was determined in patients with HR-MDS. ORR was defined by summarizing and calculating the number/percentage of patients with Complete Remission + marrow Complete Remission (CR + mCR) based on International Working Group (IWG) criteria. Based on IWG criteria CR and mCR are considered the best outcomes and used for this endpoint. CR is defined as Bone marrow (BM): ≤ 5% myeloblasts with normal maturation of all cell lines, dysplasia may persist. Peripheral Blood (PB): Hgb ≥ 11g/dL, Platelets ≥ 100 x 10^9/L, Neutrophils ≥ 1.0 x 10^9/L, Blasts 0%. mCR is defined as BM: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment. PB: if Hematologic Improvement (HI) responses, should be noted in addition to mCR (in this study, mCR absent HI is NOT considered a response). All responses must last ≥ 4 weeks. Patients who have any response will be permitted to continue treatment until relapse or progression of disease. Results are summarized using basic descriptive statistics.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 6 patients who comprised the Primary Outcome analysis were part of the HR-MDS cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 6
Participants | 4

15. Post Hoc Outcome: Best Overall Response in Patients With HR-MDS
Description: Best Overall Response was determined for patients with HR-MDS. The number/percentage of patients with Complete Remission (CR), marrow Complete Remission (mCR), and No Response is summarized based on IWG criteria. The summary also includes the number/percentage of patients who demonstrated Complete Remission with incomplete hematologic recovery (CRi).
Time Frame: At the time of censoring of data, up to ~21 months
Population: 6 patients who comprised the Primary Outcome analysis were part of the HR-MDS cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 6
Participants
  CR | 3
  mCR | 1
  CRi | 2
  No Response | 0

16. Post Hoc Outcome: Duration of Response (DOR) in AML Patients
Description: Median DOR was determined for AML patients who comprised the Primary Outcome Measure analysis. DOR was evaluated from the time of response after 12 weeks of induction until disease progression.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 21 patients who comprised the Primary Outcome analysis were part of the AML cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 21
months | 5.5 [3.9 to NA] — An upper limit for the 95% Confidence Interval for DOR was unable to be reached due to some AML patients continuing to respond to treatment at the time of cutoff for data analysis (i.e., ~21 months).

17. Post Hoc Outcome: Duration of Response (DOR) in HR-MDS Patients
Description: Median DOR was determined for HR-MDS patients who comprised the Primary Outcome Measure analysis. DOR was evaluated from the time of response after 12 weeks of induction until disease progression.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 6 patients who comprised the Primary Outcome analysis were part of the HR-MDS cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 6
months | 5.2 [4.8 to NA] — An upper limit for the 95% Confidence Interval for DOR was unable to be reached due to some HR-MDS patients continuing to respond to treatment at the time of cutoff for data analysis (i.e., ~21 months).

18. Post Hoc Outcome: Mortality
Description: Mortality at 8 weeks was assessed for the 31 patients who were evaluated as part of the Primary Outcome Measure
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 31
Participants | 0

19. Post Hoc Outcome: Measurable Residual Disease (MRD) in AML Patients Analyzed by ITT
Description: The number/percentage of AML patients analyzed by ITT who achieved Measurable Residual Disease (MRD) negativity was determined by multiparameter flow cytometry (MFC). Achieving MRD negativity after achieving remission in a cancer treatment is associated is associated with longer remissions, potentially longer survival rates, and a lower risk of relapse.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 21 patients who comprised the Primary Outcome analysis were part of the AML cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 21
Participants | 9

20. Post Hoc Outcome: Measurable Residual Disease (MRD) in AML Patients Analyzed by ITT-PP
Description: The number/percentage of AML patients analyzed by ITT-PP who achieved Measurable Residual Disease (MRD) negativity was determined by multiparameter flow cytometry (MFC). Achieving MRD negativity after achieving remission in a cancer treatment is associated is associated with longer remissions, potentially longer survival rates, and a lower risk of relapse.
Time Frame: At the time of censoring of data, up to ~21 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 19
Participants | 9

21. Post Hoc Outcome: Measurable Residual Disease (MRD) in HR-MDS Patients
Description: The number/percentage of HR-MDS patients achieving Measurable Residual Disease (MRD) negativity was determined by multiparameter flow cytometry (MFC). Achieving MRD negativity after achieving remission in a cancer treatment is associated is associated with longer remissions, potentially longer survival rates, and a lower risk of relapse.
Time Frame: At the time of censoring of data, up to ~21 months
Population: 6 patients who comprised the Primary Outcome analysis were part of the HR-MDS cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Venetoclax (Single Arm)
Number analyzed (Participants) | 6
Participants | 4

ADVERSE EVENTS:
Time Frame: All adverse events that occur on or after day 1 of cycle 1 through 30 days after the final dose of study drug (end of treatment) will be reported, up to approximately 24 months total.
Arm/Group | Decitabine/Venetoclax (Single Arm)
All-Cause Mortality (participants affected / at risk) | 4/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 28/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine/Venetoclax (Single Arm) (N=31)
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 13
Dizziness (Nervous system disorders) | 3
Weakness (General disorders) | 4 — Verbatim Tem
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Acute Kidney Injury (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 — Verbatim Term
Edema limbs (General disorders) | 1 — Verbatim Term: Peripheral edema
Peripheral Neuropathy (Nervous system disorders) | 2 — Nonspecific
Headache (Nervous system disorders) | 2
Pain (General disorders) | 3 — Verbatim Term: Pain, other
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 — Verbatim Term: Night Sweats
Decreased Appetite (Metabolism and nutrition disorders) | 5 — Verbatim Term
Creatinine Increased (Investigations) | 9 — Verbatim Term: Creatinine Elevation
Alanine aminotransferase (ALT) increased (Investigations) | 13 — Verbatim Term: ALT Elevation
Aspartate aminotransferase (AST) increased (Investigations) | 8 — Verbatim Term: AST Elevation
Blood Bilirubin Increased (Investigations) | 13 — Verbatim Term: Bilirubin Elevation
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 — Verbatim Term: Neutropenic Fever
Fever (General disorders) | 3 — Verbatim Term: Fever, non-neutropenic
Bone Marrow Hypocellular (Blood and lymphatic system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 5 — Verbatim Term: Pneumonia
Bacteremia (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 3 — Verbatim Term: Cellulitis
Urinary Tract Infection (Infections and infestations) | 4
COVID-19 (Infections and infestations) | 4 — Verbatim Term. Outcome
Respiratory Syncytial Virus (RSV) (Infections and infestations) | 2 — Verbatim Term. Outcome
Norovirus (Infections and infestations) | 1 — Verbatim Term. Outcome
Sinusitis (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT05184842/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05184842/ICF_001.pdf